CLINICAL TRIAL: NCT00523380
Title: An Open-Label Phase 2 Trial of Pegylated Liposomal Doxorubicin and rIL-21 in Ovarian Cancer Patients With Persistent or Progressive Disease After, or Relapse Within One Year of, Completion of Standard First Line Therapy
Brief Title: Efficacy Study of Recombinant Interleukin-21 in the Treatment of Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN028-1802; 2007-001506-25 (EudraCT Number)
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Cancer; Ovarian Cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: recombinant interleukin-21; Drug: caelyx (pegylated liposomal doxorubicin)

INTERVENTIONS:
Drug: recombinant interleukin-21 — Administered i.v. in treatment cycles of 28 days.
  Other Names: rIL-21; NN028
Drug: caelyx (pegylated liposomal doxorubicin) — Administered i.v. in treatment cycles of 28 days.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the efficacy of rIL-21 and Caelyx in cancer patients who have relapsed after, or have persistent disease after, first line therapy. Patients will be treated for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Advanced epithelial Ovarian Cancer (stage IIB-IV)
* Persistent or progressive disease after or relapse within one year of completion of first line therapy
* Measurable or assessable disease
* Eastern Cooperative Oncology Group status less than or equal to 2

Exclusion Criteria:

* History of any other active malignancy
* Signs of CNS metastasis
* More than one prior chemotherapy regimen
* Radiotherapy (bone) less than 4 weeks prior to start of treatment and radiotherapy (visceral) less than 8 weeks
* First line chemotherapy completed at least 1 month prior to start of treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10-04 (Actual); Primary Completion 2009-01-07 (Actual); Study Completion 2009-01-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment assessed by overall response rate (RR). RR measured and recorded using imaging techniques, CA-125 blood samples and pelvic examination. | after max. 6 treatment cycles

SECONDARY OUTCOMES:
Pharmacokinetics | Initially
IL-21 antibody formation | For the duration of the trial
Progression free survival | For the duration of the trial
Patient reported outcomes | For the duration of the trial
Biomarker assessments CA-125 | For the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (7):
- France (4):
  - Novo Nordisk Investigational Site, Lyon
  - Novo Nordisk Investigational Site, Marseille
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Villejuif
- Germany (3):
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Marburg
  - Novo Nordisk Investigational Site, Wiesbaden

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com